CLINICAL TRIAL: NCT03564249
Title: A Feasibility Study to Measure Gut Transit in Paediatric Constipation Using Novel Mini-capsules and Magnetic Resonance Imaging
Brief Title: Magnetic Resonance Imaging in Paediatric Constipation
Acronym: MAGIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14GA014
Record Dates: First submitted 2018-03-14; First posted 2018-06-20 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 Young patients with constipation (Experimental): 25 young patients that present at secondary or tertiary care with intractable constipation. They will undergo the new MRI gastrointestinal transit test (MiniCap) once before standard treatment for constipation and once after the treatment.
  Interventions: Device: MiniCap
- Group 2 Healthy participants (Experimental): 25 young healthy controls matched for gender. They will undergo the new MRI gastrointestinal transit test (MiniCap) once.
  Interventions: Device: MiniCap

INTERVENTIONS:
Device: MiniCap — The MiniCap device consists of small, completely inert mini-capsules that, once ingested, can be imaged inside the gastrointestinal tract using MRI, thereby creating a new MRI alternative to the radiopaque marker X-ray test to measure gut transit. The MRI mini- capsules are visualised in the gut using a single fat, water, in-phase and out-of-phase scan

SUMMARY:
Constipation in children is a common problem. Managing these children is difficult, partly because they do not respond to laxatives and partly because their bowel problem cannot be defined. A "gut transit time" test can add information to help choose the best therapy but this is often not carried out because of the unsuitable radiation dose involved in the current methods such as X-ray. A new Magnetic Resonance Imaging (MRI) method to measure gut transit time using inert mini-capsules, the size of small pine nuts, has recently been developed.

This study is the first feasibility test of the new mini-capsules in paediatric constipation. 25 patients and 25 healthy controls will participate. The study will measure gut transit time using MRI and the mini-capsules before and after the young patients receive standard treatment.

DETAILED DESCRIPTION:
One in ten children worldwide has constipation and it becomes chronic in 30% of these children, affecting their and their families' well-being. Managing these children is difficult, partly because they do not respond to laxatives and partly because their bowel problem cannot be defined. If the doctors could send the children for a quick test that indicates the time that food takes to travel through the gut (the "gut transit time"), they could use this information to help choose the best therapy, for example to decide if a patient needs surgery. The test could also be used to follow up the effects of different treatments. Gut transit time is often not tested due to the unsuitable radiation dose involved in the current methods such as X-ray. Doctors' decisions have to rely mostly on symptoms, leading to repeated appointments, frustration and a waste of NHS money.

A new method to measure gut transit time using mini-capsules, the size of small pine nuts, has recently been developed. The mini-capsules are swallowed but do not dissolve and their journey through the gut is imaged using Magnetic Resonance Imaging (MRI). From the images doctors can determine the gut transit time. MRI is harmless and can be used repeatedly to follow up the response to treatment.

This study will test these new mini-capsules to determine their suitability for paediatric use. Areas of interest are ease of imaging in the gut using MRI and whether they are small enough such that their emptying from the stomach and transit through the gut are similar to food. The study will test the mini-capsules in children with constipation, to measure gut transit time before and after they receive their usual treatment from their doctors. This will assess if the mini-capsules can detect changes in treatment and will make them clinically useful.

ELIGIBILITY:
Inclusion Criteria:

* Aged 7 - 18 years old
* Male or female
* Able to give assent or have a parent able to give informed consent
* Willing to allow their GP or consultant, if appropriate, to be notified of participation in the clinical investigation
* Presenting with intractable constipation at secondary or tertiary care and considered for possible treatment which may include new drugs or procedures (Group1 only)
* Healthy bowel habit and does not suffer from constipation or diarrhoea (Group 2 only)

Exclusion Criteria:

* Female participants who are pregnant, lactating or planning pregnancy during the course of the investigation.
* Any history of gastrointestinal surgery such as colectomy or small bowel resection.
* Existing ACE procedure before the first MRI scan (Group 1 only)
* Significant renal or hepatic impairment
* Contraindications for MRI scanning such as metallic implants and penetrating eye injury.
* Inability to lie flat and relatively still for less than 5 minutes
* Poor understanding of English language
* Any other significant disease or disorder (other than intractable constipation for Group 1)
* Participation in another research clinical investigation involving an investigational product in the past 12 weeks.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Whole gut transit time (hours) | 1 week time frame
  Whole gut transit time measured from the number of MiniCap retained in the bowel as detected by MRI imaging

SECONDARY OUTCOMES:
EQ-5D-Y questionnaires | Recorded at 2 time points before and after intervention (one week time frame)
  The EuroQOL five dimensions questionnaire for young (EQ-5D-Y) is the EuroQuol descriptive system for children and adolescents. It describes 5 dimensions of Quality of Life: mobility, looking after myself, doing usual activities, having pain or discomfort and feeling worried, sad or unhappy. Each dimension has 3 levels: no problems, some problems and a lot of problems. The younger patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the younger patient's health state. An EQ-5D health state is the set of responses to the 5 dimensions of EQ-5D, as completed by a patient or respondent. For instance, a fairly healthy person may have an EQ-5D health state of 1-2-1-1-1. The higher the digits the worse the health state.
EQ-VAS | Measured at 10 time points before and after intervention (one week time frame)
  The EuroQOL visual analogue scale (EQ-VAS) records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'. The scale is numbered from 1 to 100 with 100 being the best health and 0 the worst health.
AC-QoL questionnaire (total score) | Measured at 2 time points before and after intervention (one week time frame)
  The Adult carers quality of life (AC-QoL questionnaire) is a questionnaire for use with adult carers that measures quality of life in eight separate domains: support for caring; caring choice; caring stress; money matters; personal growth; sense of value; ability to care; and carer satisfaction. The questions are designed for scoring between 0 to 3 (from never to always). The composite score reflects the overall quality of life with low scores 0-40 representing a low reported quality of life and greater than 81 a high reported quality of life.
Change in whole gut transit time (hours) | Measured at 2 time points before and after standard treatment for constipation (approximately 6 months time frame)
  Change in whole gut transit time measured from the number of MiniCap retained in the bowel as detected by MRI imaging before and after standard treatment for constipation
Number of participants completing the study | Measured at 1 time point after starting the intervention (one week time frame)
  The number of participants completing the entire study will be used to assess feasibility
Number of adverse events | Measured at 1 time point after starting the intervention (one week time frame)
  The number of adverse events will be used to assess safety

CONTACTS AND LOCATIONS:
Overall Officials: Pauline H Taylor, Study Director — Nottingham University Hospitals NHS Trust
Locations (1):
- Nottingham Digestive Diseases Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided